CLINICAL TRIAL: NCT02069197
Title: Evaluation of Efficacy and Safety of Ketogenic Diet Treatment of Obesity With Co-morbid Type 2 Diabetes Mellitus and/or Obstructive Sleep Apnea.
Brief Title: Ketogenic Diet Treatment of Obesity With Co-morbid Type 2 Diabetes Mellitus and/or Obstructive Sleep Apnea
Acronym: KGDobesity
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mid-Atlantic Epilepsy and Sleep Center, LLC (Other)
Responsible Party: Principal Investigator, Pavel Klein, MD, Mid-Atlantic Epilepsy and Sleep Center, LLC
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: maes 004
Record Dates: First submitted 2013-07-19; First posted 2014-02-24 (Estimated); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Obesity; Diabetes; Obstructive Sleep Apnea
Keywords: ketogenic diet; obesity; diabetes; obstructive sleep apnea
MeSH Terms: conditions — Obesity; Diabetes Mellitus; Sleep Apnea, Obstructive | interventions — Diet, Ketogenic; Diet, Protein-Restricted; Diet, Carbohydrate-Restricted; Orlistat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ketogenic diet, lifestyle counseling (Active Comparator): ketogenic diet consisted of 3:1[fat]:[protein+carbohydrate] weight ratio with 1600kcal restriction.
  Interventions: Other: Ketogenic diet
- Orlistat, Lifestyle counseling (Active Comparator): Orlistat 120 mg TID, standardized diet and lifestyle-modification counseling based on the LEARN (Life, Exercise, Attitudes, Relationships,and Nutrition) program with recommended caloric goal of 1600 kcal/day.
  Interventions: Drug: Orlistat
- Standartized diet, Lifestyle counseling (Active Comparator): Standardized diet and lifestyle-modification counseling based on the LEARN (Lifestyle, Exercise, Attitudes, Relationship, Nutrition) program with recommended caloric goal of 1600kcal/day.
  Interventions: Other: Standardized diet

INTERVENTIONS:
Other: Ketogenic diet — ketogenic diet will consist of 3:1[fat]:[protein+carbohydrate]weight ratio with 1600 kcal restriction. Diet will last 9 months.
  Other Names: high fat, low protein, low carbohydrate diet
  Arms: Ketogenic diet, lifestyle counseling
Drug: Orlistat — Orlistat 120 mg TID for 9 months; life style intervention with recommended caloric goal of 1600 kcal/day.
  Other Names: tetrahydrolipstatin
  Arms: Orlistat, Lifestyle counseling
Other: Standardized diet — Standardized diet treatment for 9 months with recommended caloric goal of 1600kcal/day.
  Arms: Standartized diet, Lifestyle counseling

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety of ketogenic diet (KD) treatment of (i) obesity, (ii) type 2 diabetes mellitus and (iii) obstructive sleep apnea (OSA) in patients with obesity and Type 2 DM and in patients with obesity and/or OSA. This will be a randomized, open-label three arm controlled study comparing weight loss in obese participants with type 2 diabetes and/or obstructive sleep apnea treated for 9 months with 3:1 [fat]:[protein+carbohydrate] ratio, 1600 kcal/day diet (Group A) with weight loss in participants treated with orlistat 120 mg TID and lifestyle intervention consisting of dietary advice, recommended caloric goal of 1600 kcal/day (Group B), and in participants treated with only lifestyle intervention consisting of dietary advice, recommended caloric goal of 1600 kcal/day (Group C).

DETAILED DESCRIPTION:
The study sample will be randomized into three treatment arms, KD (Group A, n=50), Orlistat 120 mg TID (Group B, n=50) and dietary and lifestyle counseling (Group C, n=50) in a 1:1:1 ratio. Each arm will include 100% participants with obesity and co-morbid type 2 DM and 50% participants with co-morbid OSA. Randomization will be stratified for diabetic status.

ELIGIBILITY:
Inclusion Criteria:

* age 18-70
* ability and willingness to signed informed consent form
* BMI more than 30kg/m2, with type 2 DM and/or OSA
* For diabetic participants, stable hypoglycemic medications for at least 2 months
* For participants with OSA, previously documented polysomnogram with apnea/hypopnea index (AHI)>15/h.

Exclusion Criteria:

* BMI change of +/- 3.0 kg/m2 of baseline BMI within past 12 months.
* History of bariatric surgery ≤ 3 years prior to enrollment.
* Any systemic illness or unstable medical condition that might pose additional risk, including: cardiac, unstable metabolic or endocrine disturbances, renal or liver disease, past history of renal calculi, hyperuricemia, hypercalcemia, mitochondrial disease, known disorder of fatty acid metabolism, porphyria, and active systemic cancer.
* History of uncontrolled hyperlipidemia
* For participants with DM, change in the dose or type of hypoglycemic treatment within 2 months prior to enrollment.
* Psychosis within six months of enrollment, evidenced by treatment with anti-psychotic medications with recent medication initiation or dose increase.
* Active drug or alcohol dependence or any other factors that, in the opinion of the site investigators would interfere with adherence to study requirements;
* History of hyperthyroidism
* History of glaucoma
* History of cerebrovascular disease or unstable heart disease within 6 months of enrollment
* Pregnancy
* Use of any investigational drugs within 3 months of enrollment.
* Inability or unwillingness of subject to give written informed consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2014-01; Primary Completion 2020-08 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Change of body mass index from baseline in 9 months period | 9 months
  The change of weight and the BMI(body mass index) will be calculated.

SECONDARY OUTCOMES:
Change from baseline in glucose blood level in patients with diabetes mellitus in 9 months. | 9 months
  HbA1C, fasting serum glucose insulin and leptin levels and fasting lipid levels
Change of apnea/hypopnea index in patients with obstructive sleep apnea in patients with obesity | 9 months
  For participants with OSA, secondary outcome will include polysomnogram-derived apnea/hypopnea index.
  Level of alertness will be evaluated with Epworth Sleepiness Scale.
To evaluate safety of ketogenic diet as a treatment of obesity. | 9 months
  Evaluate in serum levels of beta-hydroxybutyrate, glucose, electrolytes, renal and liver functions, uric acid, HbA1C, serum lipid profile, insulin and leptin levels, CRP.

CONTACTS AND LOCATIONS:
Overall Officials: Pavel Klein, M.D., Principal Investigator — Mid-Atlantic Epilepsy and Sleep center
Locations (1):
- Mid-Atlantic Epilepsy and Sleep Center, LLC, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided